CLINICAL TRIAL: NCT01083381
Title: The Effect of MS14 in Association With Risperidone in Treatment of Schizophrenia: A Double Blind Randomized Control Trial
Brief Title: Is MS14 Helpful in Schizophrenia?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Farzan Institute (Other)
Responsible Party: Gholamreza Habibi, Farzan Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09123272376
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia treatment MS14 randomized clinical trial
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment group (Active Comparator): The treatment group receives Risperidone 2 mg per day in the beginning which is increased by 1 mg every day until reaching 4 mg/day; this regimen will be continued for three months. MS14 will be administered at an oral dose of 25-50 mg/kg/day in two divided doses for three months.
  Interventions: Drug: MS14; Drug: Risperidone
- Control group (Placebo Comparator): Receives the same dosage of Risperidone. Placebo is given to this group in same form and appearance as MS14 in the other arm of the study.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: MS14 — MS14 will be administered at an oral dose of 25-50 mg/kg/day in two divided doses for three months
  Arms: treatment group
Drug: Risperidone — The treatment group receives Risperidone 2 mg per day in the beginning which is increased by 1 mg every day until reaching 4 mg/day; this regimen will be continued for three months.

SUMMARY:
In this study we want to find out whether MS14 - a herbal drug- can help Schizophrenia patients or not.

DETAILED DESCRIPTION:
Schizophrenia is a chronic illness characterized by disturbances in cognition, affect and behavior, all of which have a bizarre aspect. It is a common disorder, with a prevalence of about 1%. It has an equal prevalence in both sexes although men manifest their symptoms earlier than women. [1, 2] Individuals with schizophrenia have a 2-3 fold increase in mortality rate compared to the general population. This rate had increased in recent decades. [3, 4] Most patients are incapable of maintaining their jobs and relationships. About half attempt suicide, and about 10% succeed. Most suicides occur early in the course of the illness. [1] Optimal management of schizophrenia requires psychological, social, and occupational therapies. [2] There are a lot of antipsychotic drugs which are necessary for treatment. Risperidone, an atypical antipsychotic, has been approved by the Food and Drug Administration for the treatment of schizophrenia in the adolescent population in the adolescent population. [5] Although atypical antipsychotic agents have improved outcomes in schizophrenia, their clinical potential remains limited by patients' nonadherence to medication. [6] Some of the patients with schizophrenia do not respond completely to treatment and only experience a partial improvement and remain functionally impaired. While medication has been found to be effective for the treatment of "positive" symptoms of the disease, treatment of the "negative symptoms" of schizophrenia (including lack of energy, motivation, and emotions) has historically not been very successful. [4, 5] MS14 is an Iranian herbal-marine compound that has been patented by invention and patent registration office of Islamic Republic of Iran (no: 29350) and classified as equivalent to food with no observable adverse effect level (NOAEL). [8, 9] According to analytic data this compound contains many inorganic salts or complexes and also trace elements such as bromine (Br), strontium (Sr), vanadium (V), titanium (Ti), nickel (Ni) and zinc (Zn). [10] Safety of MS14 has been confirmed by sub-acute toxicity studies in rats (clinical, histopathological, hematological and biochemical). [8] A study of MS14 in experimental allergic encephalomyelitis (EAE) model has shown that oral treatment of the EAE mice with MS14 not only halts the progression of the disease but also attenuates the inflammation in CNS indicating that this herbal-marine compound has anti-inflammatory effects [11].

Overall, alleviation of clinical and neurological symptoms in EAE mice by MS14 explained the beneficial effects of traditionally used MS14 in MS patients, an effect which could also be investigated in other groups of psychological and neurological diseases. Additionally, there are anecdotal but unconfirmed reports for the effectiveness of MS14 in patients with schizophrenia. In this regard, we have decided to perform a randomized placebo-controlled study on the effect of MS14 on schizophrenia, to assess the safety and efficacy of this compound.

ELIGIBILITY:
Inclusion Criteria:

* No other concurrent diseases
* Signing the consent form by either the patient or their guardian
* Proved diagnosis of schizophrenia through SCID structured interview

Exclusion criteria:

* Patients with treatment resistance schizophrenia
* Recent resistance to risperidone
* Contraindications of MS14 or risperidone administration
* Patients with residual or simple schizophrenia
* Age over 65 or under 18 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-10 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
response rate | after the completion of three months of therapy

SECONDARY OUTCOMES:
CGI and PANSS questionnaires as well as a questionnaire designed for drug induced side effects will be filled weekly | During the first six weeks of therapy, patients will be interviewed every week

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Vahid Shariat, Principal Investigator — Department of Psychiatry and Mental Health Research Center, Iran University of Medical Sciences
Locations (1):
- Iran Psychiatric Training and Treatment Center, Tehran, Tehran Province, Iran